CLINICAL TRIAL: NCT00531895
Title: An Open Trial of Duloxetine on Comorbid Major Depression and Chronic Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kraepelin Psiquiatria Clinica (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O021
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2007-08

CONDITIONS: Major Depression; Chronic Primary Headache
Keywords: major depression; chronic headache; antidepressant; duloxetine
MeSH Terms: conditions — Depressive Disorder, Major; Headache Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: duloxetine — duloxetine 60 mg/d
  Other Names: Cymbalta

SUMMARY:
Background: Although major depression and chronic headache are strongly associated, there is insufficient evidence on the use of antidepressants for this specific comorbidity. This trial aimed to investigate the efficiency and tolerability of duloxetine for this indication.

Methods: Thirty outpatients of our clinic, with DSM-IV major depression and concurrent primary chronic headache (chronic migraine, chronic tension-type headache or both), 18-55 years, were recruited from April 2006 to March 2007, if they scored >21 on the Montgomery-Äsberg Depression Scale (MADRS) and had no other significant clinical condition. Subjects received duloxetine 60 mg/day for 8 weeks. MADRS scores and a visual analog pain scale (VAS) were the co-primary outcome measures. WHO quality of life scale (WHOQoL BREF) scores and headache days/week were secondary outcome measures.Conclusion: In this preliminary open trial, duloxetine 60 mg/day was effective, fast acting and well tolerated for the treatment of comorbid major depression and chronic headache.

ELIGIBILITY:
Inclusion Criteria:

* Major depression (according to DSM-IV criteria)
* MADRS scores superior to 21
* Subjects meeting the International Headache Society criteria for chronic primary headache (IHSC-2 codes 1.5.1, 1.6.1, 2.3.1, 2.3.2 and 2.4.3) (ICHS, 2003)

Exclusion Criteria:

* Over 50% reduction on MADRS scores during wash-out period
* Illicit drug or alcohol dependence
* History of multiple allergies or hypersensitivity to duloxetine
* History of epilepsy or significant neurological disorder
* Significant suicide risk
* Pregnancy or lactation
* Sexually active female subjects not using an efficient contraceptive method
* Significant laboratory abnormalities at baseline
* Significant clinical disease
* Subjects meeting DSM-IV criteria for somatisation disorder. (300.81) or presenting with delusional pain symptoms.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Montgomery-Äsberg Depression Scale (MADRS) | 8 weeks
Visual Analog Scale for pain (VAS) | 8 weeks

SECONDARY OUTCOMES:
WHO Quality of Life Scale (WHOQOL BREF) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando M Volpe, MD, PhD, Principal Investigator — Hospital SOCOR
Locations (1):
- Hospital SOCOR, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Volpe FM. An 8-week, open-label trial of duloxetine for comorbid major depressive disorder and chronic headache. J Clin Psychiatry. 2008 Sep;69(9):1449-54. doi: 10.4088/jcp.v69n0912. PMID 19193344